CLINICAL TRIAL: NCT00774228
Title: Clinical Evaluation of the I-ZIP® Ocular Bandage as a Protective Ocular Bandage in Subjects Undergoing Clear Corneal Cataract Surgery With IOL Implantation: A Pivotal Study
Brief Title: I-ZIP Ocular Bandage Pivotal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITX-08-002
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Cataract
Keywords: Cataract or intraocular lens placement surgery
MeSH Terms: conditions — Cataract

ARMS (2):
- I-ZIP Ocular Bandage (Experimental): I-Zip bandage application
  Interventions: Device: I-ZIP Ocular Bandage
- Oasis 24 hour Soft Shield Collagen Corneal Shield (Active Comparator): Oasis shield application
  Interventions: Device: Oasis 24 Hour Soft Shield Collagen Corneal Shield

INTERVENTIONS:
Device: I-ZIP Ocular Bandage
  Arms: I-ZIP Ocular Bandage
Device: Oasis 24 Hour Soft Shield Collagen Corneal Shield
  Arms: Oasis 24 hour Soft Shield Collagen Corneal Shield

SUMMARY:
To evaluate the safety and performance of the I-ZIP Ocular Bandage in subjects undergoing uneventful unilateral clear corneal phacoemulsification with foldable monofocal intraocular lens (IOL) implantation compared with the Oasis 24-hour Soft Shield Collagen Corneal Shield (Oasis Medical, Inc. Glendora, California) for providing ocular protection and relief of pain or discomfort in the acute post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a cataract and is expected to undergo unilateral clear corneal cataract surgery with phacoemulsification and implantation of a posterior chamber monofocal intraocular lens through an incision ≤ 3.5mm in width measured after IOL implantation using internal calipers.

Exclusion Criteria:

* Any intraocular inflammation in the study eye that was present during the screening slit-lamp examination or presence of ocular pain in the operative eye as rated on the pre-operative NRPS
* Previous surgery (laser or incisional) or ocular trauma to the operative eye or planned multiple procedures during cataract/IOL implantation surgery
* Potential BCVA in fellow eye worse than 20/40 as assessed by the clinical Investigator
* Active or history of chronic or recurrent inflammatory eye disease (iritis, scleritis, uveitis, iridocyclitis, rubeosis iritis), evidence of acute external ocular infections, intraocular infection, dysthyroid ophthalmopathy, nasolacrimal duct obstruction, active chalazion, uncontrolled blepharitis, uncontrolled and clinically significant dry eye syndrome, anything more than trace guttata (>10 guttae in the central 6 mm of cornea), evidence of glaucoma/glaucoma suspect, corneal dystrophy or other ocular disease that would interfere with study evaluations
* Subject is currently receiving antineoplastic therapy
* Use of topical ocular steroids within 14 days and/or systemic steroids (excluding inhalants) within 30 days prior to surgery.
* Subject is an insulin-dependent diabetic or has background diabetic retinopathy (BDR), proliferative diabetic retinopathy (PDR) or compromised macular function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Device remains localized over corneal incision | 24 hours post operative

SECONDARY OUTCOMES:
Adverse ocular events | 30 days post operative

CONTACTS AND LOCATIONS:
Locations (1):
- I-Therapeutix, Inc., Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Product is not commercially available and has been discontinued

REFERENCES:
- [Derived] Dell SJ, Hovanesian JA, Raizman MB, Crandall AS, Doane J, Snyder M, Masket S, Lane S, Fram N; Ocular Bandage Study Group. Randomized comparison of postoperative use of hydrogel ocular bandage and collagen corneal shield for wound protection and patient tolerability after cataract surgery. J Cataract Refract Surg. 2011 Jan;37(1):113-21. doi: 10.1016/j.jcrs.2010.11.001. PMID 21183106